CLINICAL TRIAL: NCT05061810
Title: The Effect of a Smartphone Application Self-management Programme on Clinical Health Outcomes in Patients With Chronic Obstructive Pulmonary Disease: A Randomised Trial
Brief Title: The Effect of a Smartphone Application Self-management Programme on Clinical Health Outcomes in Patients With Chronic Obstructive Pulmonary Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Tallaght University Hospital (Other)
Responsible Party: Principal Investigator, Lisa Glynn, Respiratory Advanced Nurse Practitioner and PhD candidate, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 00017
Record Dates: First submitted 2021-07-15; First posted 2021-09-30 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: A single centre feasibility three-arm parallel randomised control trial (RCT) study. The trial consists of three groups which are, Group A, Arm 1 (standard respiratory outpatient care with a smartphone app self-management programme with follow up monthly phone calls), Group B, Arm 2 (standard respiratory outpatient care with a smartphone app and Group C, control group (standard respiratory outpatient care).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Block randomisation sequence generation (allocation ratio of 1:1:1) to ensure equilibrium between the groups. Allocation concealment will be achieved through the use of an independent healthcare provider (HCP) who will retain the random allocation sequence
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Arm 1 (Experimental): Arm 1, group A will receive standard respiratory outpatient care such as routine virtual visits to the respiratory clinic at 6 and 12 months along with the use of a smartphone app self-management programme with follow up monthly phone calls. They will be asked to use the spirobank spirometer (measures lung function, FEVI), pulse oximeter (measures oxygen saturations, SP02) and input the dyspnoea score (m MRC), step count and view the educational videos on the app twice a week for twelve months. The smartphone app self-management programme will prompt the patient once a week to remind them to input their data. Furthermore, they will receive motivational messages weekly via the app. At the routine visits they will complete questionnaires on engagement, quality of life, m MRC scale and self-efficacy at these visits over the phone. They will inform the research team of self-reported GP visits or hospital admissions due to an exacerbation of COPD.
  Interventions: Behavioral: Smartphone application self-management programme
- Group B: Arm 2 (Experimental): Those allocated to the intervention groups B will receive standard respiratory outpatient care such as routine virtual visits at 6 and 12 months to the respiratory outpatient clinic along with the use of a smartphone app self-management programme. They will be asked to use the spirobank spirometer (measures lung function, FEV1), pulse oximeter (measures oxygen saturations, SP02) and input the dyspnoea score (m MRC), their step count and view the educational videos on the app twice a week for twelve months. The smartphone app self-management programme will prompt the patient once a week to remind them to input their data. Furthermore, they will receive motivational messages weekly via the app. At the routine visits they will complete questionnaires on engagement, quality of life, m MRC scale and self-efficacy at these visits over the phone. They will inform the research team of self-reported GP visits or hospital admissions due to an exacerbation of COPD.
  Interventions: Behavioral: Smartphone application self-management programme
- Group C: Arm 3 Control group (Active Comparator): Participants in group C the control group will receive standard outpatient respiratory care which involves attending the routine visits as outlined above and informing the research team of an GP visits and or hospital admissions relating to an exacerbation of COPD. They will complete questionnaires on quality of life, m MRC scale and self-efficacy at these visits over the phone.
  Interventions: Behavioral: Smartphone application self-management programme

INTERVENTIONS:
Behavioral: Smartphone application self-management programme — The intervention in this trial is a self-management programme via a smartphone app. This self-management programme measures lung function (FEV1), oxygen saturation (SP02), dyspnoea score (m MRC) and step count. It also provides educational videos such as recognising symptoms of an exacerbation and physical activity. The smartphone app self-management programme will provide real time data monitoring resulting in baseline trends in patient's disease pattern. Additionally, it also provides subjective data that will allow the clinician to develop an understanding of the patient's quality of life.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) has a significant impact on one's quality and quantity of life resulting in increased morbidity and mortality. In Ireland, COPD has the highest hospital admissions in comparison to other countries within the organisation for economic cooperation and development (OECD). There is a need to improve knowledge and self-management behaviour in order to improve recognition of early signs of an exacerbation thereby seeking early treatment from the general practitioner (GP) thus reducing hospital admissions among this cohort . There are limited studies pertaining to the use of a comprehensive self-management programme via a smartphone app for people with COPD on a longitudinal basis.The aim of this study is to investigate the effectiveness of a smartphone application self-management programme on clinical health outcomes in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years of age
* Confirmed COPD diagnosis defined as the presence of post- bronchodilator FEV1/FVC <0.70.
* COPD category GOLD A, B, C & D.
* Those who are able to give informed consent
* Has a smart phone and is capable of using a smartphone app to input data?
* Good dexterity to use the spirometer and pulse oximeter

Exclusion Criteria:

* n/a

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this trial will measure the number of COPD exacerbations reviewed in general practice and hospital setting | 12 months
  The number of COPD self-reported exacerbations reviewed by the GP versus the hospital. COPD exacerbations are defined as an acute event described by a worsening of the patient's respiratory symptoms that is beyond normal day-to-day variations and leads to a change in medications (GOLD 2020). The primary outcome will be assessed by the research team at, three, six and twelve months using a patient self-reported approach.

SECONDARY OUTCOMES:
Engagement with technology | 12 months
  Engagement defined as a psychological state that embraces the dynamic and interactive relationship with a principal agent or object (e.g., a brand, product, or smartphone app) that satisfies the instrumental (utility) and pragmatic (emotional satisfaction) values of a consumer (Bowden 2009, Brodie et al. 2011). This outcome will be assessed by the research team at 3, 6 and 12 months using the, user engagement scale short form (O'Brien et al. 2018). This scale consists of 12 questions which the researcher will ask the participant to strongly agree-4/agree-3/disagree-2/strongly disagree-1. The overall engagement score will be calculated by adding all of the answers together and dividing by 12. The higher score indicates high levels of engagement.
Physical activity levels | 12 months
  Defined as a planned, structured, repetitive and aims to improve or maintain one or more components of physical fitness (WHO 2018). This will be measured by viewing the step count activity patient reported exercise behaviour. This outcome will be measured by the research team at 6 and 12 months
Health -related quality of life | 12 months
  • Health -related quality of life defined as "an individual's or group's perceived physical and mental health over time" (CDC 2000). This will be measured using the clinical COPD questionnaire. This questionnaire consists of 12 questions to which the participant can answer- never-0, hardly ever-1,a few times-2, several times-3, many times-4, a great many times-5, almost all of the time-6. Items are scored on a likert scale range from 0-60. The final score is the sum of all items divided by 10. Higher scores indicate a worse health status (poor quality of life).
Self-efficacy | 12 months
  Self-efficacy is defined as one's own belief in their capability to complete tasks to reach their goals (Abedi et al. 2013). This will be measured using the self-efficacy to manage chronic disease scale is made up of 6-items ranging from1 (not at all confident)-10(totally confident). The score for each item is added up. Higher number indicates higher self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Eddie Moloney, MD, Study Chair — Tallaght University Hospital
Locations (1):
- Tallaght University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Glynn L, Moloney E, Lane S, McNally E, Buckley C, McCann M, McCabe C. A Smartphone App Self-Management Program for Chronic Obstructive Pulmonary Disease: Randomized Controlled Trial of Clinical Outcomes. JMIR Mhealth Uhealth. 2025 Apr 23;13:e56318. doi: 10.2196/56318. PMID 40267465